CLINICAL TRIAL: NCT00051662
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study to Determine the Safety, Efficacy and Pharmacokinetics of Efalizumab in Subjects With Psoriatic Arthritis
Brief Title: Safety, Efficacy and Pharmacokinetics of an Antibody for Psoriatic Arthritis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: XOMA (US) LLC (Industry)
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: HUPA600
Record Dates: First submitted 2003-01-14; First posted 2003-01-16 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-09

CONDITIONS: Psoriatic Arthritis
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — efalizumab

INTERVENTIONS:
Drug: efalizumab

SUMMARY:
The purpose of this study is to determine whether a humanized monoclonal antibody (efalizumab) is safe and effective in the treatment of psoriatic arthritis (PsA)

DETAILED DESCRIPTION:
A phase II, randomized, double-blind, placebo-controlled study to:

1. Demonstrate the clinical efficacy of efalizumab in the treatment of subjects with psoriatic arthritis (PsA).
2. Evaluate the safety, tolerability and pharmacokinetics of efalizumab in the treatment of subjects with PsA

ELIGIBILITY:
Inclusion criteria:

* Diagnosed with PsA as defined by:

  * Presence of psoriasis with at least one 2 cm plaque AND
  * One of the five functional classifications of PsA
* Functional Class I, II, or III as defined by the ACR Classification of Functional Status in Rheumatoid Arthritis
* Moderate to severe disease, defined as follows:

  * At least 3 tender and 3 swollen joints (78 joint count for tenderness and 76 joints for swelling; AND
  * Either ESR ≥ 28 mm/hr, CRP ≥ 1.5 mg/dL, or morning stiffness for ≥ 30 minutes.
* Currently taking at least one of the following systemic therapies for PsA: pre-existing stable doses of NSAIDs, corticosteroids (≤ 10 mg/day), and either sulfasalazine (≤ 3 gm/day) or methotrexate (≥ 7.5 and ≤ 30 mg/week) but not both.
* 18 to 80 years of age.
* Body weight ≤ 125 kg (275 lbs).
* Candidate for systemic immunomodulatory therapy.
* Using an acceptable method of birth control.
* If female, must have a negative serum pregnancy test during screening period, must be surgically sterile, or must be at least five years postmenopausal.
* Informed about the study and signed an informed consent prior to performance of any study-related procedure.

Exclusion criteria:

* Previous treatment with efalizumab.
* Rheumatoid Factor positive without dactylitis or positive X-rays of the hands or feet, or with rheumatoid nodules.
* History of joint replacement surgery within 60 days prior to the start of study drug dosing.
* Joint replacement therapy planned within nine months subsequent to the start of study drug dosing.
* Intra-articular cortisone injections within 28 days prior to the start of study drug dosing.
* Pregnancy or lactation.
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies. Respiratory distress (dyspnea, oxygen desaturation with pO2 < 90% or onset of acute respiratory distress syndrome), flank or back pain, and/or hypotension may be signs of anaphylaxis.
* Active bacterial, viral, fungal, mycobacterium tuberculosis or atypical mycobacterium infection.
* Positive PPD test unless subject with positive PPD test completed a course of treatment for tuberculosis
* History of any opportunistic infection.
* History of a malignancy within the past five years. Subjects with a history of fully resolved, resected, basal or squamous cell carcinoma may be enrolled.
* Received any vaccine within 28 days prior to the start of study drug dosing.
* Chronic disorders apart from PsA affecting the joints, such as systemic lupus erythematosus, rheumatoid arthritis, gout, scleroderma or known reactive arthritis (e.g., Reiter's syndrome).
* COPD, asthma, or other pulmonary disease requiring more therapy than using one inhaler 4× daily.
* Failed to respond or maintain response to Enbrel.
* Received any DMARD other than methotrexate or sulfasalazine during the 28 days prior to the start of study drug dosing.
* Approved biologic PsA therapy during the 28 days or seven half-lives of the drug prior to the start of study drug dosing, whichever is the greater length of time; Enbrel within 42 days prior to the start of study drug dosing.
* Investigational drug and/or treatment during the 28 days or 7 half-lives of the drug prior to the start of study drug dosing, whichever is the greater length of time.
* Any condition which, in the opinion of the Investigator, would jeopardize the subject's safety following exposure to efalizumab.
* Liver disease (e.g., hepatitis, cirrhosis) or abnormal hepatic function (AST or ALT ≥ 2.5

  * ULN).
* Serum creatinine level ≥ 1.5 mg/dL
* Platelet count ≤ 125,000 cells/mm3
* WBC count ≤ 3,500 cells/mm3
* Total lymphocyte count ≤ 1000 cells/mm3
* Seropositive for hepatitis B
* Seropositive for hepatitis C antibody
* Seropositive for HIV
* Antinuclear antibodies titer ≥ 1:80
* History of inflammatory bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45
Dates: Study Completion 2004-02